CLINICAL TRIAL: NCT04721262
Title: Evaluation of Hyperfine Low Field Strength Portable Point-of-Care Magnetic Resonance Imaging System in Patients Receiving Ferumoxytol Infusions
Brief Title: Ferumoxytol Enhanced Hyperfine Low Field Strength MRI
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Joel M. Stein, MD, PhD, Assistant Professor of Radiology, University of Pennsylvania
Other Study IDs: 842634
Record Dates: First submitted 2020-11-02; First posted 2021-01-22 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Anemia, Hemolytic
Keywords: Anemia; Infusion; Ferumoxytol; Feraheme
MeSH Terms: conditions — Anemia, Hemolytic; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients prescribed Ferumoxytol for iron deficiency anemia: Patients with iron deficiency anemia are commonly prescribed Ferumoxytol periodically as part of their standard clinical care. Multiple studies have characterized the efficacy and safety of Ferumoxytol in the treatment of iron deficiency anemia. Patients prescribed Ferumoxytol for iron-deficiency anemia typically include otherwise healthy women with heavy menstrual periods, patients with inflammatory bowel disease, and patients with chronic kidney disease. Such patients make ideal candidates for characterizing the effects of Ferumoxytol on novel imaging devices by obviating a medically unnecessary injection of the contrast agent.
  Interventions: Device: Hyperfine Portable MRI

INTERVENTIONS:
Device: Hyperfine Portable MRI — The Hyperfine device is a newly developed MRI unit that has multiple potential advantages over standard CT or MRI including portability, easier upkeep, open design, and ease of use. Unlike CT, the Hyperfine device does not use moving parts or X-rays to generate images. Unlike routine MRI, the Hyperfine device uses two permanent magnets with open space between and around them, rather than a super-cooled superconducting magnetic tube. In contrast to CT and routine MRI, the device can be wheeled from place to place and moved into position with the patient remaining on a gurney or hospital bed. Relative to routine MRI, the device uses a very low magnetic field strength of 64 mT compared to 1.5 T or 3 T, making it safer for patients or environments with medical devices having metallic components.

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility of using Ferumoxytol as a contrast agent on a low field strength, portable magnetic resonance imaging (MRI) system. Participants receiving Ferumoxytol as part of routine clinical care for iron deficiency anemia will be recruited and scanned on the Hyperfine MRI system before and after their clinically scheduled intravenous infusion. Resultant images will be compared to assess signal intensity changes generated by the presence of Feromoxytol.

DETAILED DESCRIPTION:
Ferumoxytol is a superparamagnetic iron oxide nanoparticle (SPION) preparation that was originally designed as an MRI contrast agent, but later received FDA approval as a treatment for iron deficiency anemia. Contrast agents alter MR images by changing tissue magnetic relaxation constants such as T1 and T2 (or T2*). Gadolinium-based contrast agents decrease T1 values, causing increased signal on T1-weighted images. At low field strength, T1 values are already very short so a further decrease may provide little contrast. At typical field strengths, Ferumoxytol strongly decreases T1 and also T2 (and T2*) values, increasing signal on T1-weighted images and (conversely) decreasing signal on T2-weighted images. This T2-based contrast mechanism may be maintained at lower field strength.

Patients with iron deficiency anemia are commonly prescribed Ferumoxytol periodically as part of their standard clinical care. Multiple studies have characterized the efficacy and safety of Ferumoxytol in the treatment of iron deficiency anemia. Patients prescribed Ferumoxytol for iron-deficiency anemia typically include otherwise healthy women with heavy menstrual periods, patients with inflammatory bowel disease, and patients with chronic kidney disease. Such patients make ideal candidates for characterizing the effects of Ferumoxytol on novel imaging devices by obviating a medically unnecessary injection of the contrast agent.

Contrast agents play a key role in diagnosing and managing numerous diseases. Ferumoxytol has been used to image a variety of pathologies and organs, including tumors and inflammation in the brain, liver, pancreas, and prostate. In addition to the different magnetic relaxation properties described above, Ferumoxytol has a higher molecular weight and prolonged blood pool period compared to typical gadolinium-based agents, facilitating imaging vasculature prior to the contrast agent leaking into the extravascular tissue. This has been exploited at higher field strengths and may be particularly advantageous for low field imaging that requires longer scan times. Ferumoxytol iron particles are taken up through the reticuloendothelial system and added to physiologic iron stores, rather than being excreted through the kidneys, resulting in increased plasma half-life while also avoiding concerns related to impaired renal function that sometimes arise with other contrast agents.

The Hyperfine device is a newly developed MRI unit that has multiple potential advantages over standard CT or MRI including portability, easier upkeep, open design, and ease of use. Unlike CT, the Hyperfine device does not use moving parts or X-rays to generate images. Unlike routine MRI, the Hyperfine device uses two permanent magnets with open space between and around them, rather than a super-cooled superconducting magnetic tube. In contrast to CT and routine MRI, the device can be wheeled from place to place and moved into position with the patient remaining on a gurney or hospital bed. Relative to routine MRI, the device uses a very low magnetic field strength of 64 mT compared to 1.5 T or 3 T, making it safer for patients or environments with medical devices having metallic components.

Standard images of different types are obtained on the Hyperfine device at the push of a button on an attached touch pad. Imaging protocols include those for anatomical depiction such as balance steady-state free precession (bSFFP), T1-weighted (T1W) gradient echo (GRE), and fast low-angle shot (FLASH) as well as imaging methods focused on the detection of pathology and tissue damage such as diffusion-weighted imaging (DWI), fluid attenuated inversion recovery (FLAIR), and T2-weighted (T2W) fast spin echo (FSE). However, it is not known if existing contrast agents can provide effective contrast in the Hyperfine low-field MRI.

Thus, the primary purpose of this study is to evaluate the efficacy of Ferumoxytol as a contrast agent in low-field MRI scanners. Patients who are already receiving Ferumoxytol as a treatment for iron deficiency anemia will be scanned before and after Ferumoxytol infusion. Degree of contrast enhancement in intravascular and extravascular compartments including the cerebral vasculature and the brain parenchyma will be the primary end-point for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Prescribed Ferumoxytol for iron deficiency anemia
* Informed consent obtained from patient or a legally authorized representative

Exclusion Criteria:

1. Contraindications to routine 1.5 T MRI evaluation, including:

   * Electrical implants such as cardiac pacemakers or perfusion pumps
   * Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts or heart valves with steel parts, metal fragments, shrapnel, tattoos near the eye, steel implants, or other irremovable ferromagnetic objects
   * History of uncontrolled seizures
   * Claustrophobia
   * Weight greater than or equal to 400 lbs (181.4 kg)
2. Pregnancy
3. Inability or suspected inability to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred from the Hematology Oncology Department, scheduled to receive an intravenous infusion of Ferumoxytol as part of their standard of care (SOC) treatment for iron deficiency anemia will receive one Hyperfine MRI scan of the brain prior to their infusion and one Hyperfine MRI scan of the brain after their infusion.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Contrast enhancement | 2 thirty-five minute scans
  Changes in MRI signal intensity (contrast enhancement) produced by the presence of the Ferumoxytol contrast agent will be quantified by co-registering brain MRI studies obtained before and after administration of Ferumoxytol and determining the ratio of signal intensity values between the two sets of images (post-Ferumoxytol/pre-Ferumoxytol) in regions of interest placed separately over brain parenchyma or vascular structures. Based on the magnetic properties of Ferumoxytol, this contrast ratio is expected to be greater than one for T1-weighted scans and less than one for T2- or T2*-weighted scans.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States